CLINICAL TRIAL: NCT06734819
Title: Effectiveness of Digital Storytelling in Increasing Living Kidney Donor Recruitment in Canada
Brief Title: Storytelling to Promote Living Donor Kidney Transplant
Acronym: LDKT Stories
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Houston Methodist Transplant & Surgery Center of Excellence (Unknown)
Responsible Party: Principal Investigator, Meghan He, Principal Investigator, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: H23-02077
Record Dates: First submitted 2024-12-07; First posted 2024-12-16 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: Living Donor Kidney Transplantation; Health Equity; Patient Education; Narrative Medicine
Keywords: Living Donor Kidney Transplantation; Health Equity; Patient Education; Narrative Medicine; Digital Storytelling
MeSH Terms: conditions — Narrative Medicine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Active Comparator): Standard of care patient education materials
  Interventions: Behavioral: Standard Patient Education
- Experimental (Experimental): 2 storytelling videos in addition to standard of care patient education materials
  Interventions: Behavioral: Storytelling Video; Behavioral: Standard Patient Education

INTERVENTIONS:
Behavioral: Storytelling Video — The Living Donation Storytelling Project (LDSP) is an online video library of living donation first-person narratives aiming to inspire more people to consider LDKT (https://livingdonationstories.org/).17 As of 2020, the library has 118 stories from living donors and kidney recipients sharing their experiences with the pursuit, challenges and outcomes of transplant.18,19 Four videos were selected from the LDSP and edited to standardized duration and thematic content. Videos were cut to three minutes in length and covered the topics of 1) challenges faced when seeking LDKT, 2) life after LDKT and 3) advice for other patients considering LDKT.
  Other Names: Living Donor Storytelling Library; LDSP
  Arms: Experimental
Behavioral: Standard Patient Education — Standard of care patient education materials include verbal didactic offered during the surgical consult and pamphlets produced by Vancouver Coastal Health.

SUMMARY:
This study will examine the effectiveness of first-person storytelling in encouraging patients with end-stage renal disease to pursue Living Donor Kidney Transplant (LDKT). The Living Donation Storytelling Library LDSP is a library of videos from donors and recipients sharing their transplant stories, serving as a narrative-based transplant education resource. This study will investigate if exposure to the LDSP changes patient readiness and motivation to pursue LDKT to ultimately increase the number of donor inquiries and donor evaluations. This study will also test if the LDSP serves as a health-literate and culturally safe education approach that can effectively support racialized communities who have a disproportionately higher need for LDKT.

DETAILED DESCRIPTION:
Background: In Canada, racialized communities are 50 to 75 percent less likely to be referred for living donor kidney transplant (LDKT), identify donors, complete evaluation, and receive transplant in comparison to white patients. Several narrative-based transplant education interventions have proven to be effective in increasing LDKT pursuit among Black patients in America. However, these education interventions are labour- and time-intensive and fail to reach the general public outside the location of transplant education. Efficacy of interpersonal education interventions have also yet to be evaluated in Canadian minority populations, predominantly comprised of South Asian, East Asian and Indigenous communities.

Objective: The aim of this study is to examine the effectiveness of a narrative-based LKDT education intervention, the Living Donation Storytelling Library, in increasing transplant knowledge, health literacy, and recruitment of living donors. Secondarily, this study aims to compare hereterogeneity in viewer responses across race and gender to identify potential targeted narrative interventions for LKDT education.

Method: Two-arm randomized control trial with 80 prospective living donor kidney transplant recipients at Vancouver General Hospital in collaboration with Houston Methodist Hospital and Weill Cornell Medical Center.

ELIGIBILITY:
Inclusion Criteria:

* Waitlisted and newly referred kidney transplant candidates at the Vancouver Kidney Transplant Program
* 18 years of age or older
* Able to provide informed consent
* English literate

Exclusion Criteria:

* Inability to understand English and provide informed consent
* Transplant candidates excluded from transplantation based on clinical criteria or other contraindications for transplant
* Unwilling to disclose information on race or ethnicity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-12 (Estimated); Primary Completion 2025-08 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Readiness and Motivation | Baseline + 1 month post-intervention
  Elucidate if allowing waitlisted transplant patients to watch two videos from the LDSP will increase their motivation in pursuing LDKT. This was assessed using the validated Decisional Balance Scale measuring perceived pros and cons of pursuing LDKT. Following the prompt, "How important is this statement to your decision about living donor transplant?" was a set of 6 perceived benefits of LDKT (eg, "With a living donor transplant, I will be able to contribute to my family and friends sooner") and 6 perceived disadvantages (eg, "I don't want to involve anyone else in my health problems"). Answer choices were "1: not important," "2: slightly important," "3: important," "4: very important," "5: extremely important." Total attitude scores were calculated by subtracting the sum of perceived disadvantage scores from the sum of perceived advantage scores to obtain a range from -30 (most negative attitude towards LDKT) to +30 (most positive attitude towards LDKT).
Transplant Actions | Baseline + 1 month post-intervention
  Elucidate if allowing waitlisted transplant patients to watch two videos from the LDSP will change their actions towards pursuing LDKT. Pro-transplant behaviors were assessed using the validated Stage of Change Scale. Seven actions related to the pursuit of LDKT were listed (eg, "generally talk to people about my interest in transplant," "ask a potential donor directly to be tested"), and participants were asked if they "1: don't plan on doing this," "2: plan on doing this," or "3: already done this." Scores were calculated by summing survey responses to obtain a range from 0 (least number of actions completed in the pursuit of LDKT) to 21 (most number of actions completed in the pursuit of LDKT).

SECONDARY OUTCOMES:
Donor Inquiries and evaluations | 3 months
  Examine if allowing waitlisted transplant patients to watch two videos from the LDSP will increase the number of donor inquiries and donor evaluations.

OTHER OUTCOMES:
Health literacy and cultural safety | Immediately post-intervention
  Test if the LDSP serves as a health-literate and culturally safe education approach that can effectively support racialized communities in pursuing LDKT.
  Perceived cultural safety, health literacy accessibility, and impact of the storytelling videos were assessed using 7 prompts (eg, "After viewing the video, I feel less alone in my transplant pathway") with answer choices "1: strongly disagree," "2: disagree," "3: neutral," "4: agree," "5: strongly agree." Following survey completion, participants were invited to elaborate on their responses in an open-ended response section.
Transplant knowledge | Baseline
  Knowledge related to LDKT was assessed using the validated KART 2.0 Transplant Knowledge Subscale. This subscale is comprised of 16-question multiple choice questions regarding basic facts about LDKT (eg, "Compared to transplants from donors who have died, how long do transplants from living donors last?"). In our study, wording of some questions were modified to reflect the local healthcare system context. Scores were calculated by summing the number of correct responses to obtain a range from 0 (lowest LDKT knowledge) to 16 (highest LDKT knowledge).

CONTACTS AND LOCATIONS:
Locations (1):
- Vancouver General Hospital, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No
No personally identifiable information will be collected on participants as the data will be unidentified, and no sensitive information will be collected.

REFERENCES:
- [Result] McQueen A, Kreuter MW, Kalesan B, Alcaraz KI. Understanding narrative effects: the impact of breast cancer survivor stories on message processing, attitudes, and beliefs among African American women. Health Psychol. 2011 Nov;30(6):674-82. doi: 10.1037/a0025395. Epub 2011 Sep 5. PMID 21895370
- [Result] Waterman AD, Nair D, Purnajo I, Cavanaugh KL, Mittman BS, Peipert JD. The Knowledge Assessment of Renal Transplantation (KART) 2.0: Development and Validation of CKD and Transplant Knowledge Scales. Clin J Am Soc Nephrol. 2022 Apr;17(4):555-564. doi: 10.2215/CJN.11490821. Epub 2022 Mar 24. PMID 35332061
- [Result] Davis L, Iraheta YA, Ho EW, Murillo AL, Feinsinger A, Waterman AD. Living Kidney Donation Stories and Advice Shared Through a Digital Storytelling Library: A Qualitative Thematic Analysis. Kidney Med. 2022 May 21;4(7):100486. doi: 10.1016/j.xkme.2022.100486. eCollection 2022 Jul. PMID 35755303
- [Result] Wood EH, Waterman AD, Pines R. Storytelling to Inspire Dialysis Patients to Learn about Living Donor Kidney Transplant. Blood Purif. 2021;50(4-5):655-661. doi: 10.1159/000512651. Epub 2021 Jan 13. PMID 33440381
- [Result] Waterman AD, Wood EH, Ranasinghe ON, Faye Lipsey A, Anderson C, Balliet W, Holland-Carter L, Maurer S, Aurora Posadas Salas M. A Digital Library for Increasing Awareness About Living Donor Kidney Transplants: Formative Study. JMIR Form Res. 2020 Jul 21;4(7):e17441. doi: 10.2196/17441. PMID 32480362
- [Result] Boulware LE, Hill-Briggs F, Kraus ES, Melancon JK, Senga M, Evans KE, Troll MU, Ephraim P, Jaar BG, Myers DI, McGuire R, Falcone B, Bonhage B, Powe NR. Identifying and addressing barriers to African American and non-African American families' discussions about preemptive living related kidney transplantation. Prog Transplant. 2011 Jun;21(2):97-104; quiz 105. doi: 10.1177/152692481102100203. PMID 21736237
- [Result] Waterman AD, Davis LA, Al Awadhi S. Unraveling Barriers in Access to Living Donor Kidney Transplantation for South Asian Canadian Populations. Am J Kidney Dis. 2024 Jun;83(6):710-712. doi: 10.1053/j.ajkd.2024.01.519. Epub 2024 Apr 11. No abstract available. PMID 38613542
- [Result] Lui E, Gill J, Hamid M, Wen C, Singh N, Okoh P, Xu X, Boakye P, James CE, Waterman AD, Edwards B, Mucsi I. Racialized and Immigrant Status and the Pursuit of Living Donor Kidney Transplant - a Canadian Cohort Study. Kidney Int Rep. 2024 Feb 1;9(4):960-972. doi: 10.1016/j.ekir.2024.01.044. eCollection 2024 Apr. PMID 38765593
- [Result] Purnell TS, Hall YN, Boulware LE. Understanding and overcoming barriers to living kidney donation among racial and ethnic minorities in the United States. Adv Chronic Kidney Dis. 2012 Jul;19(4):244-51. doi: 10.1053/j.ackd.2012.01.008. PMID 22732044
- [Result] Hamid M, Gill J, Okoh P, Yanga N, Gupta V, Zhang JC, Singh N, Matelski J, Boakye P, James CE, Waterman A, Mucsi I. Knowledge About Renal Transplantation Among African, Caribbean, and Black Canadian Patients With Advanced Kidney Failure. Kidney Int Rep. 2023 Sep 22;8(12):2569-2579. doi: 10.1016/j.ekir.2023.09.018. eCollection 2023 Dec. PMID 38106596
- [Result] Alsahafi M, Leung L, Partovi N, Yee J, Yoshida EM. Racial differences between solid organ transplant donors and recipients in British Columbia 2005-2009: a follow-up study since the last analysis in 1993-1997. Transplantation. 2013 Jun 15;95(11):e70-1. doi: 10.1097/TP.0b013e3182928261. No abstract available. PMID 23732288
- [Result] de Groot IB, Veen JI, van der Boog PJ, van Dijk S, Stiggelbout AM, Marang-van de Mheen PJ; PARTNER-study group. Difference in quality of life, fatigue and societal participation between living and deceased donor kidney transplant recipients. Clin Transplant. 2013 Jul-Aug;27(4):E415-23. doi: 10.1111/ctr.12165. Epub 2013 Jun 30. PMID 23808752

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-03-07): https://cdn.clinicaltrials.gov/large-docs/19/NCT06734819/Prot_SAP_000.pdf
  • Informed Consent Form (2024-03-07): https://cdn.clinicaltrials.gov/large-docs/19/NCT06734819/ICF_001.pdf